CLINICAL TRIAL: NCT04995887
Title: RUBY: Treating Abnormal Postpartum Uterine Bleeding or Postpartum Hemorrhage With the Jada® System - A Post-Market Registry
Brief Title: RUBY Post-Market Registry on the Jada® System
Acronym: RUBY
Status: Completed | Type: Observational
Sponsor: Alydia Health (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-05 v1.0; Protocol No. PPH-05 (Other: Alydia Health)
Record Dates: First submitted 2021-07-13; First posted 2021-08-09 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Postpartum Hemorrhage
Keywords: Vacuum-Induced Hemorrhage-Control (VHC); Jada; Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- C-Section Delivery with EBL ≥ 1500 mL: Patients with ≥ 1500 mL estimated blood loss (EBL) at time of Jada insertion for cesarean delivery; data collection will continue until a minimum of 100 patients are enrolled in each group/category or until March 31, 2022 (whichever occurs first).
  Interventions: Device: Jada® System
- C-Section Delivery with EBL < 1500 mL: Patients with < 1500 mL EBL at time of Jada insertion for cesarean delivery; data collection will continue until a minimum of 100 patients are enrolled in each group/category or until March 31, 2022 (whichever occurs first).
  Interventions: Device: Jada® System
- Vaginal Delivery with EBL ≥ 1000 mL: Patients with ≥ 1000 mL EBL at time of Jada insertion for vaginal delivery; data collection will continue until a minimum of 100 patients are enrolled in each group/category or until March 31, 2022 (whichever occurs first).
  Interventions: Device: Jada® System
- Vaginal Delivery with EBL < 1000 mL: Patients with < 1000 mL EBL at time of Jada insertion for vaginal delivery; data collection will continue until a minimum of 100 patients are enrolled in each group/category or until March 31, 2022 (whichever occurs first).
  Interventions: Device: Jada® System

INTERVENTIONS:
Device: Jada® System — The Jada® System is intended to provide control and treatment of abnormal postpartum uterine bleeding or hemorrhage when conservative management is warranted. It is a teardrop-shaped, soft silicone ring that is placed into the uterus, where gentle suction is applied to cause the uterus to contract and shrink in size, compressing the blood vessels so the bleeding stops.
  Other Names: Vacuum-induced Hemorrhage Control; Obstetric-Gynecologic Specialized Manual Instrument

SUMMARY:
The RUBY Study is a multicenter, observational, post-market registry designed to collect observational data on patients treated with the Jada System in the post-market setting.

DETAILED DESCRIPTION:
The purpose of this registry is to collect observational data on patients treated with the Jada System in the post-market setting. Data collection will include observations of effectiveness and safety of the device. Additional outcome data related to resource utilization will also be included.

ELIGIBILITY:
Inclusion Criteria:

• Use of the Jada System (inserted into the patient and connected to vacuum).

NOTE: There is no Exclusion Criteria in this protocol.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Conditions treated occur only in females of childbearing age (i.e., postpartum hemorrhage or abnormal postpartum uterine bleeding).
Study Population: Patients included are all identified through review of the medical charts as having received Jada treatment starting from the center's first commercial use of the Jada System. This chart review will be ongoing until the specified date or until a minimum of 100 patients are enrolled in each of the groups described below (whichever occurs first):
  1. ≥ 1500 mL estimated blood loss (EBL) at time of Jada insertion (C-S)
  2. < 1500 mL EBL at time of Jada insertion (C-S)
  3. ≥ 1000 mL EBL at time of Jada insertion (vaginal)
  4. < 1000 mL EBL at time of Jada insertion (vaginal)
  Up to a maximum of 50 sites can be included in this registry. Each IRB approval constitutes a "site."
Sampling Method: Probability Sample
Enrollment: 809 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy: Cessation of PPH | 24 hours
  Proportion of patients with atony-related abnormal postpartum uterine bleeding or PPH successfully treated with the Jada System. Treatment success is defined as the avoidance of escalated non-surgical or surgical intervention to control abnormal postpartum uterine bleeding or PPH after the Jada System was used.
  Note: Concomitant treatment with uterotonics or uterine compression sutures does not constitute escalation (i.e., failure). However, if the Jada treatment was aborted to instead administer treatment with compression sutures for ongoing bleeding, then the event does meet the escalation (i.e., failure) definition.
Safety: device-related Adverse Events | 24 hours through time of discharge.
  Rates of procedure- and device-related adverse events.

SECONDARY OUTCOMES:
Rate of non-surgical or surgical procedures other than Jada | 24 hours
  Rate of non-surgical or surgical procedures other than Jada for atony-related bleeding after Jada was used
Transfusion rates | 24 hours through time of discharge.
  Rate of blood transfusions
In-dwelling time of Jada during treatment | 24 hours
  In-dwelling time (i.e., insertion of Jada to removal of Jada)
Time spent in care settings | 24 hours through time of discharge.
  Time spent in care settings (e.g., L&D, OR, Delivery Room, Postpartum Room, ICU, Other) from Jada treatment through discharge
Length of stay | 24 hours through time of discharge.
  Length of stay (LOS) from delivery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Dena Goffman, MD, Principal Investigator — Columbia University
Locations (16):
- United States (16):
  - Loma Linda University, Loma Linda, California
  - ChristianaCare, Newark, Delaware
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Oshsner Baptist, New Orleans, Louisiana
  - Allina (Abbott Northwestern), Minneapolis, Minnesota
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai, New York, New York
  - Nyph/Cumc, New York, New York
  - University Hospitals, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Ohio Health, Gahanna, Ohio
  - UPMC - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Charleston Birth Place, Mt. Pleasant, South Carolina
  - University of Utah, Salt Lake City, Utah
  - Charleston Area Medical Center, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Gulmezoglu AM, Lawrie TA, Hezelgrave N, Oladapo OT, Souza JP, Gielen M, Lawn JE, Bahl R, Althabe F, Colaci D, Hofmeyr GJ. Interventions to Reduce Maternal and Newborn Morbidity and Mortality. In: Black RE, Laxminarayan R, Temmerman M, Walker N, editors. Reproductive, Maternal, Newborn, and Child Health: Disease Control Priorities, Third Edition (Volume 2). Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2016 Apr 5. Chapter 7. Available from http://www.ncbi.nlm.nih.gov/books/NBK361904/ PMID 27227224
- [Background] Callaghan WM, Kuklina EV, Berg CJ. Trends in postpartum hemorrhage: United States, 1994-2006. Am J Obstet Gynecol. 2010 Apr;202(4):353.e1-6. doi: 10.1016/j.ajog.2010.01.011. PMID 20350642
- [Background] Mulic-Lutvica A, Bekuretsion M, Bakos O, Axelsson O. Ultrasonic evaluation of the uterus and uterine cavity after normal, vaginal delivery. Ultrasound Obstet Gynecol. 2001 Nov;18(5):491-8. doi: 10.1046/j.0960-7692.2001.00561.x. PMID 11844171
- [Background] Andersen HF, Hopkins MP. Chapter 80: postpartum hemorrhage. In: Sciarra JJ, editor. Gynecology and obstetrics, volume 2. Philadelphia, PA: Lippincott Williams & Wilkins; 2004.
- [Background] Lyon DS. Chapter 90: postpartum care. In: Sciarra JJ, editor. Gynecology and obstetrics, volume 2. Philadelphia, PA: Lippincott Williams & Wilkins; 2004.
- [Background] Baskett TF. A flux of the reds: evolution of active management of the third stage of labour. J R Soc Med. 2000 Sep;93(9):489-93. doi: 10.1177/014107680009300913. No abstract available. PMID 11089490
- [Background] Main EK, Goffman D, Scavone BM, Low LK, Bingham D, Fontaine PL, Gorlin JB, Lagrew DC, Levy BS; National Partnership for Maternal Safety; Council on Patient Safety in Women's Health Care. National Partnership for Maternal Safety: Consensus Bundle on Obstetric Hemorrhage. Obstet Gynecol. 2015 Jul;126(1):155-62. doi: 10.1097/AOG.0000000000000869. PMID 26241269
- [Background] Goffman D, Ananth CV, Fleischer A, D'Alton M, Lavery JA, Smiley R, Zielinski K, Chazotte C; Safe Motherhood Initiative Obstetric Hemorrhage Work Group. The New York State Safe Motherhood Initiative: Early Impact of Obstetric Hemorrhage Bundle Implementation. Am J Perinatol. 2019 Nov;36(13):1344-1350. doi: 10.1055/s-0038-1676976. Epub 2019 Jan 4. PMID 30609429
- [Background] Shields LE, Smalarz K, Reffigee L, Mugg S, Burdumy TJ, Propst M. Comprehensive maternal hemorrhage protocols improve patient safety and reduce utilization of blood products. Am J Obstet Gynecol. 2011 Oct;205(4):368.e1-8. doi: 10.1016/j.ajog.2011.06.084. Epub 2011 Jun 29. PMID 22083059
- [Background] Rossen J, Okland I, Nilsen OB, Eggebo TM. Is there an increase of postpartum hemorrhage, and is severe hemorrhage associated with more frequent use of obstetric interventions? Acta Obstet Gynecol Scand. 2010 Oct;89(10):1248-55. doi: 10.3109/00016349.2010.514324. PMID 20809871
- [Background] Della Torre M, Kilpatrick SJ, Hibbard JU, Simonson L, Scott S, Koch A, Schy D, Geller SE. Assessing preventability for obstetric hemorrhage. Am J Perinatol. 2011 Dec;28(10):753-60. doi: 10.1055/s-0031-1280856. Epub 2011 Jun 22. PMID 21698554
- [Background] American College of Obstetricians and Gynecologists. ACOG Practice Bulletin: Clinical Management Guidelines for Obstetrician-Gynecologists Number 76, October 2006: postpartum hemorrhage. Obstet Gynecol. 2006 Oct;108(4):1039-47. doi: 10.1097/00006250-200610000-00046. PMID 17012482
- [Background] Zelop CM. Postpartum hemorrhage: becoming more evidence-based. Obstet Gynecol. 2011 Jan;117(1):3-5. doi: 10.1097/AOG.0b013e318202ec9a. No abstract available. PMID 21173639
- [Background] Purwosunu Y, Sarkoen W, Arulkumaran S, Segnitz J. Control of Postpartum Hemorrhage Using Vacuum-Induced Uterine Tamponade. Obstet Gynecol. 2016 Jul;128(1):33-36. doi: 10.1097/AOG.0000000000001473. PMID 27275795
- [Background] D'Alton ME, Rood KM, Smid MC, Simhan HN, Skupski DW, Subramaniam A, Gibson KS, Rosen T, Clark SM, Dudley D, Iqbal SN, Paglia MJ, Duzyj CM, Chien EK, Gibbins KJ, Wine KD, Bentum NAA, Kominiarek MA, Tuuli MG, Goffman D. Intrauterine Vacuum-Induced Hemorrhage-Control Device for Rapid Treatment of Postpartum Hemorrhage. Obstet Gynecol. 2020 Nov;136(5):882-891. doi: 10.1097/AOG.0000000000004138. PMID 32909970
- [Derived] Rood KM, Bianco A, Biggio JR, Smid MC, Simhan HN, Li J, Yong C, Carney PI, Croft DJ, Goffman D. Real-world use of a vacuum-induced hemorrhage-control device in births <34 weeks gestational age. J Matern Fetal Neonatal Med. 2025 Dec;38(1):2451658. doi: 10.1080/14767058.2025.2451658. Epub 2025 Feb 9. PMID 39924257
- [Derived] Goffman D, Rood KM, Bianco A, Biggio JR, Dietz P, Drake K, Heilman E, Hopkins M, De Four Jones M, Katz T, Martin C, Prasad M, Smid MC, Wine KD, Ryan R, Yong C, Carney PI, Simhan HN. Real-World Utilization of an Intrauterine, Vacuum-Induced, Hemorrhage-Control Device. Obstet Gynecol. 2023 Nov 1;142(5):1006-1016. doi: 10.1097/AOG.0000000000005366. Epub 2023 Sep 13. PMID 37713322